CLINICAL TRIAL: NCT02640391
Title: Predictive Factors of Endoscopic Mucosal Healing in Quiescent Ulcerative Colitis: Prospective Observational Multicenter Study
Brief Title: Predictive Factors of Endoscopic Mucosal Healing in Quiescent Ulcerative Colitis
Acronym: PINQLE
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Other Study IDs: KMU-151215
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; fecal calprotectin; mucosal healing
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Quiescent UC: Patients with quiscent UC who will undergo colonoscopy for surveillance or mucosal healing check up
  Interventions: Other: colonoscopy

INTERVENTIONS:
Other: colonoscopy
  Other Names: fecal calprotectin; fecal immunochemical test; Rome III criteria for IBS

SUMMARY:
The purpose of this study is to determine whether fecal calprotectin, fecal immunochemical test, and Rome III criteria for irritable bowel syndrome (IBS) can predict mucosal healing in patients with quiescent ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis who have no change of medication for at least 6 months
* Patients with ulcerative colitis who are in remission (Mayo score <3)
* Patients with ulcerative colitis who will undergo colonoscopy for surveillance or mucosal healing check-up

Exclusion Criteria:

* Patients who refuse to participate
* Patients who have a history of colectomy
* Patients who have instinal stricture or perforation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inactive UC (Mayo score <3) who are scheduled to undergo colonoscopy for surveillance or mucosal healing check-up
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mucosal healing | 1 week
  Endoscopic Mayo subscore <1
Fecal calprotectin | 1 week
Fecal immunochemical test | 1 week

SECONDARY OUTCOMES:
Rome III criteria for IBS | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, PhD, Principal Investigator — Keimyung University School of Medicine
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No